CLINICAL TRIAL: NCT01054781
Title: Open-labelled, Multicenter Phase II Study of Intensified 1st Cycle Rituximab Plus 8th Cycles of R-CHOP Chemotherapy in Patients With Advanced or Bulky CD20+ Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Intensified 1st Cycle Rituximab Plus 8th Cycles of R-CHOP Chemotherapy in Patients With Advanced or Bulky CD20+ Diffuse Large B-cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: WonSeog Kim , M.D., PhD., Samsung Medical Center,Division of Hematology-Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-12-005
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL)
Keywords: Diffuse Large B-Cell Lymphoma (DLBCL); rituximab; CHOP
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rituximab — 1st cycle R+R-CHOP 2-8th cycle R-CHOP

SUMMARY:
The purpose of this study is to evaluate the complete response (CR) rate after Intensified 1st cycle Rituximab plus 3rd cycles of R-CHOP in DLBCL

ELIGIBILITY:
Inclusion criteria

1. Histologically confirmed CD20 positive Diffuse Large B-cell Lymphoma (DLBCL)
2. Advanced stage: stage III, IV and/or bulky disease (largest diameter ≥ 10.0 cm) regardless of stage
3. Previously untreated.
4. Performance status: ECOG 0-2.
5. Age ≥ 18
6. At least one or more bidimensionally measurable lesion(s)

   * ≥ 2 cm by conventional CT
   * ≥ 1 cm by spiral CT
   * skin lesion (photographs should be taken) ≥ 2 cm
   * measurable lesion by physical examination ≥ 2 cm
7. Cardiac ejection fraction ≥ 50 % as measured by MUGA or 2D ECHO without clinically significant abnormalities
8. Adequate renal function: serum creatinine level < 2 mg/dL (177 μmol/L)
9. Adequate liver functions:

   * Transaminase (AST/ALT) < 3 X upper normal value (or < 5 x ULN in the presence of DLBCL involvement of the liver)
   * Bilirubin < 2 X upper normal value (or < 5 x ULN in the presence of DLBCL involvement of the liver)
10. Adequate hematological function: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL, unless abnormalities are due to bone marrow involvement by lymphoma
11. Life expectancy ≥ 6 months
12. A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are < 1 years after the onset of menopause.
13. Informed consent

Exclusion criteria

1. Other subtypes NHL than DLBCL
2. Patients who transformed follicular lymphoma or other indolent lymphoma
3. Primary Central Nervous System (CNS) DLBCL;
4. CNS involvement by lymphoma or any evidence of spinal cord compression. Brain CT/MRI is only mandatory (within 4 weeks) in case of clinical suspicion of CNS involvement by lymphoma. Patients who have only had prophylactic intrathecal chemotherapy against CNS disease are eligible.
5. Patients with a known history of HIV seropositivity or HCV (+). Patients who have HBV (+) are eligible. However, primary prophylaxis using antiviral agents (i.e. lamivudine) is recommended for HBV carrier to prevent HBV reactivation during whole treatment period.
6. Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
7. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
8. Other serious illness or medical conditions

   * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
   * History of significant neurological or psychiatric disorders including dementia or seizures
   * Active uncontrolled infection (viral, bacterial or fungal infection)
   * Other serious medical illnesses
9. Known hypersensitivity to any of the study drugs or its ingredients (i.e., hypersensitivity to Polysorbate 20, CHO cell products, or recombinant human antibodies)
10. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the complete response (CR) rate after Intensified 1st cycle Rituximab plus 3rd cycles of R-CHOP in DLBCL and | 12 months

SECONDARY OUTCOMES:
To evaluate the overall response rate of R+R-CHOP | 12 months
To evaluate the duration of overall response | 12 months
To evaluate the safety and tolerability of the R+R-CHOP combination treatment. | 12 months
To evaluate the progression free survival. | 12 months
To estimate the overall survival. | 12 months
To explore prognostic or predictive biomarkers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: WonSeog Kim, M.D., PhD., Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim YR, Kim JS, Kim WS, Eom HS, Yang DH, Bae SH, Kim HJ, Lee JH, Oh SJ, Yoon SS, Kwak JY, Choi CW, Kim MK, Oh SY, Kang HJ, Nam SH, Shim H, Park JS, Mun YC, Suh C; Korean Society of Hematology Lymphoma Working Party. Intensified First Cycle of Rituximab Plus Eight Cycles of Cyclophosphamide, Doxorubicin, Vincristine, and Prednisolone with Rituximab Chemotherapy for Advanced-Stage or Bulky Diffuse Large B-Cell Lymphoma: A Multicenter Phase II Consortium for Improving Survival of Lymphoma (CISL) Study. Cancer Res Treat. 2023 Oct;55(4):1355-1362. doi: 10.4143/crt.2023.271. Epub 2023 Mar 30. PMID 36996864